CLINICAL TRIAL: NCT05746481
Title: A Phase II Clinical Trial of Tiragolumab in Combination With Atezolizumab in Patients With Non-small Cell Lung Cancer (NSCLC) and Untreated Brain Metastases.
Brief Title: Tiragolumab and Atezolizumab in Patients With Non-squamous Non-small Cell Lung Cancer (NSCLC) and Untreated Brain Metastases
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Decision by agent provider
Sponsor: Liza Villaruz, MD (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Liza Villaruz, MD, Associate Professor of Medicine, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCC 22-045
Record Dates: First submitted 2023-02-16; First posted 2023-02-27 (Actual); Results first posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Non-small Cell Lung Cancer
Keywords: PD-L1 tumor proportion score (TPS); salvage radiation therapy; brain metastases
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Brain Neoplasms | interventions — Tiragolumab; atezolizumab; Pemetrexed; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single Treatment Arm (Experimental): Tiragolumab in combination with atezolizumab, pemetrexed, and carboplatin.
  Interventions: Drug: Tiragolumab; Drug: Atezolizumab; Drug: Pemetrexed; Drug: Carboplatin

INTERVENTIONS:
Drug: Tiragolumab — Tiragolumab (an investigational novel immune checkpoint inhibitor): 600 mg IV for induction treatment administered on Day 1 of each 21-day cycle for 4 cycles. Maintenance therapy will continue with tiragolumab on Day 1 of each 21-day cycle.
  Other Names: RO7092284
Drug: Atezolizumab — Atezolizumab (monoclonal antibody): 1200 mg IV administered on Day 1 of each 21-day cycle.
  Other Names: Tecentriq; RO5541267
Drug: Pemetrexed — Pemetrexed (antifolate antineoplastic agent chemotherapy): 500 mg/m2 administered IV on Day 1 of each 21-day cycle.
  Other Names: Alimta; Pemfexy
Drug: Carboplatin — Carboplatin AUC 5 (alkylating agent chemotherapy): injection administered on Day 1 of each 21-day cycle.
  Other Names: Paraplatin

SUMMARY:
This clinical trial is aimed at the evaluation of the safety and clinical activity of tiragolumab in combination with atezolizumab with or without chemotherapy in the first line treatment of metastatic non-squamous NSCLC patients with asymptomatic untreated brain metastases.

DETAILED DESCRIPTION:
This is a phase II clinical trial aimed at the evaluation of the safety and clinical activity of tiragolumab in combination with atezolizumab with or without chemotherapy in the first line treatment of metastatic non-squamous NSCLC patients with asymptomatic untreated brain metastases. Patients with at least one untreated evaluable brain metastasis of 5 mm or more will be enrolled. Lesions previously treated with SRS may not be used as target lesions. Patients will be required to undergo an on-treatment brain MRI at three weeks for safety purposes. Additional restaging will occur at nine-week intervals. PD-L1 tumor proportion score (TPS) will be determined utilizing an FDA-approved test by local testing.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed non-squamous NSCLC.
* In patients treated with the combination of tiragolumab and atezolizumab, patients must have PDL1 TPS >50%, as determined by an FDA-approved test.
* Patients must have asymptomatic brain metastases with at least one untreated evaluable (per RANO-BM) brain metastasis of 5 mm or more. A growing lesion previously treated with whole brain radiotherapy is acceptable given the lower incidence of radiation necrosis. Lesions previously treated with SRS may not be used as target lesions.

  o Patients are not required to have measurable disease outside the CNS per RECIST 1.1.
* Prior chemotherapy, immunotherapy or radiation given with curative intent in early stage or locoregionally advanced NSCLC is permitted, if completed more than 12 months prior to initiation of study treatment.
* Prior radiation with palliative intent in the metastatic setting to non-CNS lesions is permitted (no wash-out period).
* Age ≥18 years.
* ECOG performance status ≤ 1.
* Life expectancy ≥12 weeks.
* Patients must have normal organ and marrow function as defined below:

  * Absolute neutrophil count ≥1,500/mcL
  * Platelets ≥100,000/mcL
  * Total bilirubin ≤ institutional upper limit of normal (ULN)
  * AST(SGOT)/ALT(SGPT) ≤2.5 × institutional ULN
  * Creatinine Clearance (CrCl) ≥45 mL/min/1.73 m2
* No known history of HIV, with the following exception: patients who are HIV positive are eligible provided they are stable on anti-retroviral therapy, have a CD4 count ≥ 200/µL, and have an undetectable viral load.
* Negative hepatitis B surface antigen (HBsAg) test at screening. If positive, an HBV DNA test must also be performed to determine if the patient has an HBV infection, which would render the patient ineligible. Patients receiving treatment with anti-viral therapy for HBV are excluded.
* Negative hepatitis C antibody. If positive, an HCV RNA test must also be performed to determine if the patient has an HCV infection, which would render the patient ineligible.
* Availability of a representative tumor specimen for exploratory biomarker research.
* For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraception:
* Women must remain abstinent or use contraceptive methods with a failure rate of < 1% per year during the treatment period and for 90 days after the final dose of tiragolumab, 5 months after the final dose of atezolizumab, and 6 months after the final dose of paclitaxel, pemetrexed, gemcitabine, carboplatin, or cisplatin.

  * A woman is considered to be of childbearing potential if she is postmenarchal, has not reached a postmenopausal state (≥ 12 continuous months of amenorrhea with no identified cause other than menopause), and has not undergone surgical sterilization (i.e., removal of ovaries, fallopian tubes, and/or uterus) or another cause as determined by the investigator (e.g., Müllerian agenesis). Per this definition, a woman with a tubal ligation is considered to be of childbearing potential. The definition of childbearing potential may be adapted for alignment with local guidelines or regulations.
  * Examples of contraceptive methods with a failure rate of < 1% per year include bilateral tubal ligation, male sterilization, hormonal contraceptives that inhibit ovulation, hormone-releasing intrauterine devices, and copper intrauterine devices.
  * The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not adequate methods of contraception. If required per local guidelines or regulations, locally recognized adequate methods of contraception and information about the reliability of abstinence will be described in the local Informed Consent Form.
* Women who would like to become pregnant after study treatment discontinuation should seek advice on oocyte cryopreservation prior to initiation of study treatment because of the possibility of irreversible infertility due to treatment with cisplatin and carboplatin.
* For men: agreement to remain abstinent (refrain from heterosexual intercourse) or use a condom, and agreement to refrain from donating sperm, as defined below:

  * With a female partner of childbearing potential, men who are not surgically sterile must remain abstinent or use a condom plus an additional contraceptive method that together result in a failure rate of < 1% per year during the treatment period, for 90 days after the final dose of tiragolumab, and for 6 months after the final dose of paclitaxel, pemetrexed, gemcitabine, carboplatin or cisplatin. Men must refrain from donating sperm during this same period.
  * With a pregnant female partner, men must remain abstinent or use a condom during the treatment period for 90 days after the final dose of tiragolumab, and for 6 months after the final dose of paclitaxel, pemetrexed, gemcitabine, carboplatin, or cisplatin to avoid exposing the embryo.
  * The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not adequate methods of contraception. If required per local guidelines or regulations, locally recognized adequate methods of contraception and information about the reliability of abstinence will be described in the local Informed Consent Form.
* Men who would like to father a child after study treatment initiation should be advised regarding the conservation of sperm prior to treatment because of the possibility of irreversible infertility resulting from chemotherapies used in this study.
* Women of childbearing potential must have a negative serum pregnancy test result within 14 days prior to initiation of study treatment.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Symptoms related to brain metastases requiring CNS radiation ≤ 2 weeks of treatment initiation are exclusionary. Steroids greater than prednisone 10 mg/d or equivalent, or anti-epileptic therapy ≤ 2 weeks of treatment initiation are exclusionary.
* Prior systemic therapy for metastatic disease is not allowed.
* Patients whose tumors harbor oncogenic drivers with an approved 1st line therapy (e.g. EGFR, ALK, and ROS1 alterations) are excluded.
* Patients who are receiving any other investigational agents.
* Active or history of autoimmune disease or immune deficiency, including, but not limited to, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, antiphospholipid antibody syndrome, Wegener granulomatosis, Sjögren syndrome, Guillain-Barré syndrome, or multiple sclerosis, with the following exceptions:

  * Patients with a history of autoimmune-related hypothyroidism who are on thyroid replacement hormone are eligible for the study.
  * Patients with controlled Type 1 diabetes mellitus who are on an insulin regimen are eligible for the study.
  * Patients with eczema, psoriasis, lichen simplex chronicus, or vitiligo with dermatologic manifestations only (e.g., patients with psoriatic arthritis are excluded) are eligible for the study provided all of following conditions are met:

    * Rash must cover < 10% of body surface area
    * Disease is well controlled at baseline and requires only topical corticosteroids
  * No occurrence of acute exacerbations of the underlying condition requiring psoralen plus ultraviolet A radiation, methotrexate, retinoids, biologic agents, oral calcineurin inhibitors, or high potency or oral corticosteroids within the previous 12 months.
* History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on screening chest computed tomography (CT) scan. History of radiation pneumonitis or fibrosis in a radiation field is permitted.
* History of leptomeningeal disease.
* Active tuberculosis.
* Significant cardiovascular disease (such as New York Heart Association Class II or greater cardiac disease, myocardial infarction, or cerebrovascular accident) within 3 months prior to initiation of study treatment, unstable arrhythmia, or unstable angina.
* Major surgical procedure, other than for diagnosis, within 4 weeks prior to initiation of study treatment, or anticipation of need for a major surgical procedure during the study.
* History of malignancy other than NSCLC within 2 years prior to screening, with the exception of malignancies with a negligible risk of metastasis or death (e.g., 5-year OS rate ≥ 90%).
* Severe infection within 2 weeks prior to initiation of study treatment, including, but not limited to, hospitalization for complications of infection, bacteremia, or severe pneumonia.
* Prior allogeneic stem cell or solid organ transplantation.
* Any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding that contraindicates the use of an investigational drug, may affect the interpretation of the results, or may render the patient at high risk from treatment complications.
* Treatment with a live, attenuated vaccine within 4 weeks prior to initiation of study treatment, or anticipation of need for such a vaccine during atezolizumab treatment or within 5 months after the final dose of atezolizumab.
* Treatment with systemic immunosuppressive medication (including, but not limited to, corticosteroids in excess of prednisone 10 mg/d or equivalent, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-TNF-α agents) within 2 weeks prior to initiation of study treatment, or anticipation of need for systemic immunosuppressive medication during study treatment, with the following exceptions:

  * Patients who received acute, low-dose systemic immunosuppressant medication or a one-time pulse dose of systemic immunosuppressant medication (e.g., 48 hours of corticosteroids for a contrast allergy) are eligible for the study.
  * Patients who received mineralocorticoids (e.g., fludrocortisone), corticosteroids for chronic obstructive pulmonary disease (COPD) or asthma, or low-dose corticosteroids for orthostatic
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to atezolizumab or other agents used in study.
* History of severe allergic anaphylactic reactions to chimeric or humanized antibodies or fusion proteins.
* Known hypersensitivity to Chinese hamster ovary cell products or to any component of the atezolizumab or tiragolumab formulation.
* Pregnancy or breastfeeding, or intention of becoming pregnant during study treatment, within 90 days after the final dose of tiragolumab, 5 months after the final dose of atezolizumab, or 6 months after the final dose of pemetrexed, gemcitabine, paclitaxel, carboplatin, or cisplatin o Women of childbearing potential must have a negative serum pregnancy test result within 14 days prior to initiation of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2023-08-10 (Actual); Primary Completion 2024-08-19 (Actual); Study Completion 2025-11-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Liza C Villaruz, MD, Principal Investigator — UPMC Hillman Cancer Center
Locations (1):
- UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Single Treatment Arm
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Single Treatment Arm
Number analyzed (Participants) | 3
Age, Continuous [Mean (Full Range); unit: years] | 68.33 [56 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Rate of Initiation of Salvage Radiation Therapy to Central Nervous System (CNS)
Description: The proportion of patients that require salvage radiation therapy to the CNS (within 18 weeks from study initiation). Salvage radiation therapy is radiation treatment given for suspected recurrent malignant disease.
Time Frame: Up to 18 weeks
Population: Enrolled patients
Measure: Count of Participants; unit: Participants
Arm/Group | Single Treatment Arm
Number analyzed (Participants) | 3
Participants | 0

2. Secondary Outcome: Adverse Events Related to Treatment
Description: Adverse Events and Serious Adverse Events per Common Terminology Criteria for Adverse Events CTCAE v5.0, at least possibly related to trial treatment.
Time Frame: Up to 12 months
Measure: Number; unit: participants
Arm/Group | Single Treatment Arm
Number analyzed (Participants) | 3
participants
  Alkaline phosphatase increased | 1
  Anemia | 3
  Anorexia | 1
  Aspartate aminotransferase increased | 1
  Chronic Kidney Disease | 1
  Creatinine increased | 1
  Eczema | 2
  Edema limbs | 1
  Fatigue | 2
  Hypophosphatemia | 1
  Hypothyroidism | 1
  infusion related reaction | 1
  Lipase increased | 2
  Lung infection | 1
  Lymphocyte count decreased | 3
  Mucositis oral | 1
  non-papular rash | 1
  Platelet count decreased | 1
  Pruritus | 1
  Rash acneiform | 1
  Serum amylase increased | 1
  Sinus tachycardia | 1
  Thyroid stimulating hormone increased | 1
  White blood cell decreased | 2

3. Secondary Outcome: Brain Metastasis Response Rate (BMRR)
Description: Number of patients with brain metastases that experience a Complete or Partial Response per RANO-BM. RANO Criteria: Complete Response (CR):disappearance of all enhancing disease (measurable and non-measurable), sustained for at least 4 weeks, stable or improved non-enhancing FLAIR/T2W lesions, no new lesions; clinical features - no corticosteroids (physiological replacement doses allowed) clinically stable or improved. Partial Response (PR): 50% or more decrease of all measurable enhancing lesions sustained for at least 4 weeks no progression of non-measurable disease stable or improved non-enhancing FLAIR/T2W lesions no new lesions; clinical features stable or reduced corticosteroids (compared to baseline) clinically stable or improved. Progressive disease (PD): either one of: any new lesions at least 20% relative and 5 mm absolute increase of SOD of target lesions compared to smallest SOD ever recorded. Stable disease (SD): not meeting criteria for PD or PR.
Time Frame: Up to 24 months
Population: Treated patients.
Measure: Count of Participants; unit: Participants
Arm/Group | Single Treatment Arm
Number analyzed (Participants) | 3
Participants
  Complete Response | 0
  Partial Response | 2
  Stable Disease | 1

4. Secondary Outcome: Response Per RANO Criteria
Description: Response per RANO Criteria: Complete Response (CR):disappearance of all enhancing disease (measurable and non-measurable), sustained for at least 4 weeks, stable or improved non-enhancing FLAIR/T2W lesions, no new lesions; clinical features
  - no corticosteroids (physiological replacement doses allowed) clinically stable or improved. Partial Response (PR): 50% or more decrease of all measurable enhancing lesions sustained for at least 4 weeks no progression of nonmeasurable disease stable or improved non-enhancing FLAIR/T2W lesions no new lesions; clinical features stable or reduced corticosteroids (compared to baseline) clinically stable or improved.
Time Frame: Up to 24 months
Population: Treated patients evaluable for response.
Measure: Count of Participants; unit: Participants
Arm/Group | Single Treatment Arm
Number analyzed (Participants) | 3
Participants
  Complete Response (CR) | 0
  Partial Response (PR) | 2

5. Secondary Outcome: Response Per RECIST
Description: The proportion of participants experiencing Complete or Partial Response assessed using RECIST v1.1. Per RECIST v1.1: Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (target or nontarget) with reduction in short axis to <10 mm. Partial Response (PR): ≥30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: Up to 24 months
Population: Treated patients evaluable for radiologic response.
Measure: Count of Participants; unit: Participants
Arm/Group | Single Treatment Arm
Number analyzed (Participants) | 2
Participants
  Complete Response (CR) | 0
  Partial Response (PR) | 2

6. Secondary Outcome: Progression-free Survival (PFS) - Per Patient
Description: The length of time from start of treatment that a patient lives with disease but without disease progression. Per RECISIT v1.1: Progressive Disease (PD):≥20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). The sum must also demonstrate an absolute increase of ≥5 mm. The appearance ≥1 new lesion(s) is considered progression.
Time Frame: Up to 24 months
Population: Treated patients evaluable for response.
Measure: Number; unit: months
Arm/Group | Single Treatment Arm
Number analyzed (Participants) | 3
months
  Patient 1 | 18.8
  Patient 2 | 10.8
  Patient 3 | 13.5

7. Secondary Outcome: Overall Survival (OS)
Description: The median duration of time from start of treatment until death from any cause.
Time Frame: Up to 24 months
Population: All enrolled patients.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Single Treatment Arm
Number analyzed (Participants) | 3
months | NA [NA to NA] — Median was not reached as no event was observed in the any patients.

8. Secondary Outcome: Progression-free Survival After Initiation of Salvage XRT (PFS2)
Description: The length of time during and after treatment and after after initiation of salvage radiation therapy (XRT) that a patient lives with disease but without disease progression. Per RECISIT v1.1: Progressive Disease (PD):≥20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). The sum must also demonstrate an absolute increase of ≥5 mm. The appearance ≥1 new lesion(s) is considered progression.
Time Frame: Within 18 weeks of study initiation
Population: No patients received salvage radiation therapy to the CNS.
Arm/Group | Single Treatment Arm
Number analyzed (Participants) | 0

9. Secondary Outcome: PD-L1 Tumor Proportion Score (TPS)
Description: Tumor Proportion Score (TPS) indicates protein expression by measuring the percentage of viable tumor cells showing partial or complete membrane staining at any intensity. The specimen is considered to have PD-L1 expression if TPS ≥ 1% and high PD-L1 expression if TPS ≥ 50%.
Time Frame: Up to 24 months
Population: Treated patients who completed surgery.
Measure: Number; unit: percentage of PD-L1 positive tumor cells
Arm/Group | Single Treatment Arm
Number analyzed (Participants) | 3
percentage of PD-L1 positive tumor cells
  Patient 1 | 90
  Patient 2 | 1
  Patient 3 | 0

10. Secondary Outcome: Progression-free Survival (PFS)
Description: The median length of time from start of treatment that a patient lives with disease but without disease progression. Per RECISIT v1.1: Progressive Disease (PD):≥20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). The sum must also demonstrate an absolute increase of ≥5 mm. The appearance ≥1 new lesion(s) is considered progression.
Time Frame: Up to 24 months
Population: Treated patients evaluable for response.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Single Treatment Arm
Number analyzed (Participants) | 3
months | 13.48 [10.58 to NA] — Upper bound of 95% CI not reached due to low number of patients/events observed.

11. Secondary Outcome: Overall Survival (OS) - Per Patient
Description: The duration of time from start of treatment until death from any cause, or the last clinical follow-up.
Time Frame: Up to 24 months
Population: All enrolled patients.
Measure: Number; unit: months
Arm/Group | Single Treatment Arm
Number analyzed (Participants) | 3
months
  Patient 1 | 18.8
  Patient 2 | 10.6
  Patient 3 | 14.4

ADVERSE EVENTS:
Time Frame: Adverse Events data were collected for up to 12 months. All-Cause Mortality data was collected for up to 24 months. Per-patient Survival presented in Outcome Measure 7 is defined as "The length of time from start of treatment that patients remain still alive". No patients have had the event of death while they were on study. Participants were monitored/assessed for All-Cause Mortality for up to 24 months (while on study)
Arm/Group | Single Treatment Arm
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 1/3
Other Adverse Events (participants affected / at risk) | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Single Treatment Arm (N=3)
Stroke (Nervous system disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Single Treatment Arm (N=3)
Abdominal pain (Gastrointestinal disorders) | 1
Alanine aminotransferase increased (Investigations) | 2
Alkaline phosphatase increased (Investigations) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1
Anemia (Blood and lymphatic system disorders) | 3
Aspartate aminotransferase increased (Investigations) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1
Belching (Gastrointestinal disorders) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Bruising (Injury, poisoning and procedural complications) | 1
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1
Chills (General disorders) | 1
Chronic Kidney Disease (Renal and urinary disorders) | 1
Confusion (Psychiatric disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Creatinine increased (Investigations) | 1
Dysarthria (Nervous system disorders) | 1
Dysgeusia (Nervous system disorders) | 1
Eczema (Skin and subcutaneous tissue disorders) | 1
Edema limbs (General disorders) | 2
Eosinophilia (Blood and lymphatic system disorders) | 1
Fall (Injury, poisoning and procedural complications) | 1
Fatigue (General disorders) | 3
Fever (General disorders) | 1
Flu like symptoms (Vascular disorders) | 1
Fracture (Injury, poisoning and procedural complications) | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1
Hypercalcemia (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 3
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
Hyperkalemia (Metabolism and nutrition disorders) | 1
Hypertension (Vascular disorders) | 2
Hyponatremia (Metabolism and nutrition disorders) | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 1
Hypotension (Vascular disorders) | 1
Hypothyroidism (Endocrine disorders) | 1
infusion related reaction (Investigations) | 1
left eye flashes of light (Eye disorders) | 1
Leukocytosis (Blood and lymphatic system disorders) | 1
Lipase increased (Investigations) | 2
Lung infection (Infections and infestations) | 1
Lymphocyte count decreased (Investigations) | 2
Memory impairment (Nervous system disorders) | 1
Mucositis oral (Gastrointestinal disorders) | 1
Muscle cramp (Musculoskeletal and connective tissue disorders) | 1
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1
Muscle weakness right-sided (Nervous system disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 2
Non-cardiac chest pain (General disorders) | 1
non-papular rash (Skin and subcutaneous tissue disorders) | 1
pain - right shoulder (General disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Paresthesia (Nervous system disorders) | 2
petechial rash (hands) (Skin and subcutaneous tissue disorders) | 1
Photosensitivity (Skin and subcutaneous tissue disorders) | 1
Platelet count decreased (Investigations) | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 2
Serum amylase increased (Investigations) | 1
Sinus bradycardia (Cardiac disorders) | 1
Sinus tachycardia (Cardiac disorders) | 2
Syncope (Nervous system disorders) | 1
Thrush (Investigations) | 1
Thyroid stimulating hormone increased (Investigations) | 1
Tremor (Nervous system disorders) | 1
Weight gain (Investigations) | 1
White blood cell decreased (Investigations) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-10-16): https://cdn.clinicaltrials.gov/large-docs/81/NCT05746481/Prot_SAP_000.pdf